CLINICAL TRIAL: NCT02126696
Title: Study on Non-communicable and Selected Communicable Chronic Comorbidities Among HIV-positive Patients on Anti-retroviral Therapy in Rural Lesotho and Their Association to Virologic Outcome
Brief Title: Comorbidities and Virologic Outcome Among Patients on Anti-retroviral Therapy in Rural Lesotho
Status: Completed | Type: Observational
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Swiss Foundation for Excellence and Talent in Biomedical Research (Unknown); SolidarMed - Swiss Organization for Health in Africa (Unknown); University of Basel (Other); Central Laboratories, University Hospitals Basel-Land (Liestal) (Unknown)
Responsible Party: Sponsor
Other Study IDs: CART-1
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: HIV; Metabolic Syndrome; Depression; Alcoholism; Hepatitis
Keywords: Anti-retroviral Therapy; Lesotho; Southern Africa; Comorbidity; Virologic failure
MeSH Terms: conditions — Metabolic Syndrome; Depression; Alcoholism; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Frozen human plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients on anti-retroviral therapy: The cohort consists of patients on first-line anti-retroviral therapy since at least 6 months, followed at one of the facilities involved in the study.

SUMMARY:
This study is conducted in a cohort of HIV-positive patients on first-line anti-retroviral therapy (ART) in rural health facilities in Lesotho, Southern Africa. It examines virologic treatment failure as well as chronic communicable and non-communicable comorbidities among patients on ART. The study has two phases. Phase 1 consists of a cross-sectional survey to determine prevalence of treatment failure as well as the prevalence of the following comorbidities: diabetes mellitus, arterial hypertension, dyslipidemia, depression, alcohol use disorder, hepatitis B and hepatitis C. Phase 2 is a cohort study, where patients with treatment failure or a comorbidity or both are followed-up for 12 months.

DETAILED DESCRIPTION:
Background

Owing to successful scale-up and decentralization of anti-retroviral therapy (ART) in rural Lesotho, the number of persons infected with HIV who stay alive increased dramatically. The new situation of HIV having turned from a deadly disease into a chronic but manageable condition creates a new challenge to health care providers in rural facilities of the country. Patients on long-time ART may suffer from comorbidities endangering the success of ART and their health and/or from ART-failure due to development of resistance of the virus. The magnitude of the burden of comorbidities as well as ART- failure has not been examined extensively in Lesotho yet.

Objectives of the Study

The study has six major objectives:

1. To assess the prevalence of virologic failure and genotype-resistance of HIV among patients on ART in rural Lesotho.
2. To assess the prevalence of hepatitis C and hepatitis B among patients on ART in rural facilities in Lesotho
3. To assess the prevalence of diabetes mellitus, arterial hypertension and dyslipidaemia among patients on ART in rural facilities in Lesotho
4. To assess the prevalence of depression and alcohol use disorder among patients on ART in rural facilities in Lesotho
5. To examine associations between chronic comorbidities and virologic outcome among patients on ART in rural Lesotho
6. To follow-up patients with virologic failure and/or comorbidity(ies) among patients on ART in rural Lesotho

Design/Methods

The study is planned to take place in two districts of Lesotho: Botha-Bothe and Thaba-Tseka. Prevalence of the selected comorbidities is measured in a cross-sectional, facility-based survey in eight health centers and two hospitals from the two districts. Patients with a detectable viral load will receive enhanced adherence counselling and a second viral load measurement after 2-3 months. In case of confirmed virologic failure, a genotype resistance testing will be done before patients are switched to second-line. Patients with specific comorbidities or patients with virologic failure who had been switched to second-line ART will be followed-up in a cohort study 12-18 months after the survey.

Expected Results and Impact

Prevalence of the selected comorbidities will inform the Ministry of Health as well as its implementing partners on which chronic conditions might be most urgent to be addressed among patients on ART in Lesotho and the national HIV-programme may be used to leverage on for other chronic conditions. Data on virologic failure will inform on the prevalence of virologic failure among a previously not virologically monitored cohort. Moreover it will provide data on the resistance patterns among patients who fail on first-line ART and on the one-year outcome after switch to a second-line regimen.

ELIGIBILITY:
Inclusion Criteria:

* on anti-retroviral therapy ≥ 6 months
* informed consent given

Exclusion Criteria:

* on anti-retroviral therapy for < 6 months or documented treatment interruption of ≥ 7 days during the last 3 months
* children < 16 years without the caretaker who can provide informed consent for study participation
* patients on second-line anti-retroviral therapy

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients on anti-retroviral therapy ≥ 6 months followed at one of the facilities involved in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1754 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of comorbidities among patients on anti-retroviral therapy in rural Lesotho | at enrollment
  The prevalence of the following comorbidities/conditions will be assessed:
  * Diabetes Mellitus
  * Arterial Hypertension
  * Dyslipidemia
  * Depression
  * Alcohol use disorder
  * Hepatitis B
  * Hepatitis C
Prevalence of virologic failure and genotype resistance patterns among patients on anti-retroviral therapy who were not monitored virologically | At enrollment
  All patients on first-line ART ≥ 6 months will receive viral load testing. Those with a detectable viral load will receive enhanced adherence counselling and again a viral load measurement 3 months after the initial viral load (as recommended by the consolidated WHO-guidelines). In case of persistent virologic failure (2 times detectable viral load) a genotype resitance testing will be done and patients will be switched to second-line ART. This will allow to validate the WHO algorithm for virologic failure in a remote, resource-limited setting.

SECONDARY OUTCOMES:
1-year follow-up outcomes of patients with virologic failure and subsequent switch to second-line ART | 12-18 months after enrollment
  Patients with virologic failure at enrollment will be followed-up after 12-18 months to assess the following outcomes:
  1. clinical outcome: alive and on ART / lost to follow-up / dead
  2. virological outcome: viral load suppressed / viral load detectable
1-year outcomes of patients with comorbidities diagnosed at enrollment | 12-18 months after enrollment
  Patients diagnosed with a specific comorbidity at enrollment (see first primary outcome) will be followed-up to assess their outcome after one year:
  1. clinical outcome: alive and on ART / lost to follow-up / dead
  2. virologic outcome: viral load suppressed / viral load detectable
Predictors of sustained virologic failure 3 months after a detectable viral load at initial measurement | enrollment + 3 months
  Potential clinical/laboratory predictors to predict sustained virologic failure among patients with a detectable viral load at initial measurement will be collected at enrollment.
Association of comorbidities and virologic outcomes among patients on anti-retroviral therapy in rural Lesotho | at enrollment
  Virologic outcome of anti-retroviral therapy will be compared between patient-groups with and without one or more of the comorbidities listed under the first primary outcome.

OTHER OUTCOMES:
Association of patient-wealth and virologic failure among patients on ART in rural Lesotho | at enrollment
  Patient wealth will be assessed using the wealth index developed by the Demographic Health Survey Lesotho (http://dhsprogram.com/publications/publication-FR241-DHS-Final-Reports.cfm). Virologic outcome of patients will be stratified by wealth-quintile
Virologic outcome of patients on anti-retroviral therapy at decentralized centers as compared to patients followed at the hospitals | at enrollment
  Patients will be stratified if they were followed at a health center (nurse-led) or at a hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus D Labhardt, MD, MIH, Principal Investigator — Swiss Tropical & Public Health Institute; Christoph Hatz, Prof, Study Director — Swiss Tropical & Public Health Institute; Thomas Klimkait, Prof, Study Chair — Department of Biomedicine, University of Basel
Locations (2):
- Lesotho (2):
  - Seboche Hospital, Butha-Buthe, Butha-Buthe
  - Paray Hospital, Thaba-Tseka, Thaba-Tseka

REFERENCES:
- [Derived] Labhardt ND, Muller UF, Ringera I, Ehmer J, Motlatsi MM, Pfeiffer K, Hobbins MA, Muhairwe JA, Muser J, Hatz C. Metabolic syndrome in patients on first-line antiretroviral therapy containing zidovudine or tenofovir in rural Lesotho, Southern Africa. Trop Med Int Health. 2017 Jun;22(6):725-733. doi: 10.1111/tmi.12872. Epub 2017 May 4. PMID 28342180
- [Derived] Cerutti B, Broers B, Masetsibi M, Faturiyele O, Toti-Mokoteli L, Motlatsi M, Bader J, Klimkait T, Labhardt ND. Alcohol use and depression: link with adherence and viral suppression in adult patients on antiretroviral therapy in rural Lesotho, Southern Africa: a cross-sectional study. BMC Public Health. 2016 Sep 8;16(1):947. doi: 10.1186/s12889-016-3209-4. PMID 27608764